CLINICAL TRIAL: NCT06413329
Title: The Association Between Physical Activity Level and Post-operative Prognosis
Status: Not yet recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: K5803
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Elective Operation Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- exposure: Patients' preoperative exercise level met the standard of American Exercise guidelines.
  Interventions: Behavioral: preoperative physical activity level within 3 months
- control: Patients' preoperative exercise level did not meet the standard of American Exercise guidelines

INTERVENTIONS:
Behavioral: preoperative physical activity level within 3 months — The exercise compliance criteria are moderate exercise of at least 150 minutes per week or high-intensity exercise of at least 75 minutes per week.
  Groups: exposure

SUMMARY:
The study primarily focuses on adult patients who underwent elective surgery at Peking Union Medical College Hospital. The physical activity level before surgery within the past 3 months is the main exposure factor and postoperative quality of life score (EQ-5D-3L utility index) is the main outcome indicator. The correlation between patients' preoperative physical activity level and their surgical outcomes will be explored in this study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing elective surgery at Peking Union Medical College Hospital

Exclusion Criteria:

* 1. Patients scheduled for surgery with minimal impact on overall health (including eye surgery, abortion, hysteroscopy, conization, gastroscopy, vascular angiography, and superficial surgery, etc.) 2. Orthopedic and cardiac surgery patients 3. Patients who are unable to live independently or have significant limitations in physical activity prior to surgery 4. Patients who have difficulty communicating verbally and cannot complete the questionnaire 5. Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing elective surgery at Peking Union Medical College Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 324 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Quality of life after the surgery | two weeks, one month and three months after surgery
  EQ-5D-3L index will be collected and calculated for evaluation of patients' quality of life after the surgery

SECONDARY OUTCOMES:
postoperative hospitalization days | one week after discharge
  from surgery to discharge
ICU length of stay | one week after discharge
  ICU length of stay
postoperative complications | three months after surgery
  Complications occurring within three months after surgery

IPD SHARING:
Plan to Share IPD: No